CLINICAL TRIAL: NCT04159753
Title: An Evaluation Study of Patient Experience Comparing Tonic Vs. Burst Spinal Cord Stimulation For Chronic Pain
Brief Title: Patient Experience Comparing Tonic Vs. Burst Spinal Cord Stimulation For Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 2 patients enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael D. Osborne, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-001362
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-11

CONDITIONS: Chronic Pain
Keywords: Spinal cord stimulator (SCS)
MeSH Terms: conditions — Chronic Pain | interventions — Implantable Neurostimulators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Spinal Cord Stimulator (Other): Burst neurostimulation
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — We will record patient's experience on the 30-Day FDA approved Burst Spinal Cord Stimulator Trial (BurstDR™, Abbott Saint Jude Medical).
  Other Names: Neurostimulator

SUMMARY:
Researchers are evaluating if subjects who have already experienced tonic spinal cord stimulation would have a better pain relief status with burst spinal cord stimulation.

DETAILED DESCRIPTION:
The study is a controlled trial with subjects that have an already-implanted SCS device (Eon Mini™) and are not satisfied with their pain relief status. As part of medical standard of care, patients with already-implanted Eon family tonic implantable pulse generators (IPGs) have the opportunity to experience burst stimulation for 30-Day Trial FDA approved. The aim of the study record patients experience during the 30-Day Trial using standard questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years-old
* Diagnosed with chronic pain
* Have an already-implanted Eon Family IPG for a minimum period of 6 months
* Are interested in trying burst technology by reprograming their IPG for 2-3 weeks according to the 30-Day Trial standard of care
* Signed informed consent

Exclusion Criteria:

* Subject's overall Beck Depression Inventory II Score is >24 or has a score of 3 on question 9 relating to suicidal thoughts or wishes at the screening visit; If subjects scores indicate suicidal thoughts, subject is going to be evaluated further if they will be subjects to Baker's act
* Subject is currently receiving, applying or considering seeking disability payments, workers compensation, or is involved in disability litigation
* Subject has an infusion pump or any other implantable neurostimulator device
* Subjects with a separate, concurrent, clinically significant or disabling chronic pain problem that requires additional medical or surgical treatment
* Subject's pain originates from peripheral vascular disease
* Subject is immunocompromised
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection
* Subject has history of cancer requiring active treatment in the last 6 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in Pain scores using Numeric Rating Scale (1-10)
Pain quality, intensity and localization | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in pain perception using Short-Form McGill Pain Questionnaire-2
Pain perception | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in pain perception using the Pain Catastrophizing Scale self-reported survey

SECONDARY OUTCOMES:
Depression | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in depression scores using Beck Depression Inventory-II self reported survey
Functioning | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in patient's functioning using Oswestry Disability Index self-reported survey
Participant self-evaluation of Quality of Life | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in quality of life scores using self-reported questionnaire Short-From-36 Health Survey
Participant's impression of Quality of Life | Participants will be followed at baseline, before and after the 2-3 weeks burst reprograming trial, and 3-8 months after burst trial ends
  Change in quality of life using Patient Global Impression of Change self-reported survey on activity limitations, symptoms and emotions

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osborne, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials